CLINICAL TRIAL: NCT03928834
Title: Implementing a Sustainable Adherence Intervention and Monitoring Virologic Suppression and Drug Resistance Among HIV-infected Adolescents Receiving Antiretroviral Therapy in Zimbabwe (SAPHRA)
Brief Title: Sustainable Adherence and Prevention of HIV Drug Resistance in Adolescents
Acronym: SAPHRA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a delay in getting protocol approvals and hence the study would not be completed in time.
Sponsor: University of Zimbabwe (Other)
Collaborators: King's College London (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GH002118-01
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Medication Adherence; HIV Drug Resistance
Keywords: Adolescents; HIV drug resistance; Genotyping; Dried blood spots
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Two-arm, cluster-randomized trial
  1) clinics that provide the Standard of care (SOC)VL testing and management to adolescents and 2) clinics that provide an enhanced adherence package consisting of VL testing using Dried Blood Spots(DBS), including the Nzira Itsva ( NI) intervention and low-cost genotyping and drug resistance monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapted Nzira Itsva Intervention (Experimental): Participants will be attending clinics that provide an enhanced adherence package to the adolescents consisting of viral load (VL) testing using DBS, including the Nzira Itsva(NI) intervention and low-cost genotyping and drug resistance monitoring
  Interventions: Behavioral: Adapted Nzira Itsva
- Standard of Care( SOC) (No Intervention): Participants will be attending clinics that provide the standard of care (SOC) VL testing and management to adolescents

INTERVENTIONS:
Behavioral: Adapted Nzira Itsva — Adolescents will be provided an enhanced adherence package consisting of VL testing using DBS, including the NI intervention and low-cost genotyping and drug resistance monitoring. Participants receiving the intervention will have their first session after recruitment and enrollment, and will schedule up to 4 additional booster sessions at a time convenient for them spaced approximately 1 month apart. This may be modified after the formative assessment.
  Arms: Adapted Nzira Itsva Intervention

SUMMARY:
The overall goal of this study is to determine if implementation of a package of interventions that includes DBS-based VL monitoring, coupled with an evidence-based intervention to improve ART adherence using cognitive-behavioral principles and genotyping for those with persistent viremia decreases 12-month virologic failure rates among HIV-infected adolescents compared with standard of care (SOC).

DETAILED DESCRIPTION:
In 2014, UNAIDS set ambitious goals to achieve 90% virologic suppression rates among individuals on antiretroviral therapy (ART). In Zimbabwe, this is an ambitious target, particularly among adolescents; less than 5% of human immunodeficiency virus (HIV)-infected individuals received HIV viral load (VL) testing in 2015, as reported by Ministry of Health and Child Care in Zimbabwe and treatment failure rates among adolescents range between 25-37% (Makadzange et al., 2015). Adolescents failing ART also have high rates of drug resistance. Scalable strategies to facilitate improved VL monitoring, adherence support, and genotyping for those with persistent viremia are urgently needed. The investigators have shown that dried blood spot (DBS) samples can be used for routine VL monitoring on existing technologies (Makadzange et al., 2017) They have also adapted an evidence-based, widely-used, cognitive behavioral therapy (CBT) adherence intervention (Life-Steps) for use in Zimbabwe and have identified a low-cost genotyping strategy that can facilitate detection of drug resistance mutations (DRMs) using already existing real-time polymerase chain reaction technology. The primary study objective is to determine if implementation of a package of care that includes DBS-based VL monitoring, coupled with an evidence-based intervention to improve ART adherence using cognitive-behavioral principles as well as genotyping for individuals with persistent viremia decreases 12-month virologic failure rates among HIV-infected adolescents compared with standard of care (SOC). The investigators hypothesize that the proposed package of care will result in a decrease in virologic failure rates among adolescents. They will also adapt and integrate Nzira Itsva for Adolescents (NI), a cultural adaptation of Life-Steps, into routine care as an adherence support intervention for HIV-infected adolescents, and implement a novel, low-cost genotyping assay using Pan-Degenerate Amplification and Adaptation (PANDAA) of viral ribonucleic acid (RNA) as a point mutation assay for the detection of drug resistance in parallel with Sanger sequencing. Process and cost data will be collected for subsequent cost-analysis. The proposed intervention will be a two-arm, cluster-randomized trial in Mashonaland West and Matabeleland North provinces of Zimbabwe. The units of randomization will be public and largely rural clinics within the provinces, with sites randomized to the intervention or to the SOC. The study is anticipated to show that the use of DBS in routine monitoring of adolescents is feasible, and to show that CBT, if incorporated into routine counselling activities, can complement VL monitoring and genotyping to reduce treatment failure rates and preserve therapeutic options for infected adolescents. The results of this study will have important implications in Zimbabwe and other low-income countries in sub-Saharan Africa with a large proportion of HIV-infected adolescents. The study will include young adolescents aged 10- <14years, as well as older adolescents aged 15-19 years and therefore provide data that will guide implementation of strategies for virologic success in the growing number of perinatally-infected children who are surviving on ART into adolescence, as well as for behaviorally-infected adolescents. The study will be performed within 44 clinics in Matabeleland North and Mashonaland West provinces, and will recruit 828 adolescents. A multidisciplinary consortium with the expertise to conduct this study has been assembled. The consortium includes public health practitioners, a biostatistician, basic scientists with extensive experience in virology and development of novel technologies, HIV clinicians with experience in implementation science, global mental health, and behavioral psychology experts. The consortium will work in partnership with the Ministry of Health (MOH) to implement this protocol and ensure its success.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive adolescents aged 10-19 years who know their status
2. On ART for at least 6 months as per clinic records: the patient will have attended the clinic as shown in clinic records at least once since initiation AND will have re-filled their ART at least once since initiation as shown in clinic records..
3. Planning to stay in care at that facility for at least 12 months

Exclusion Criteria:

1. Participant and/or caregiver unable to give consent and assent
2. Those participants who the healthcare worker considers to be too ill to participate

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
To determine VL suppression rates in adolescents in SOC and intervention arm | 12 months
  Arm-specific VL suppression rates will be estimated by the proportion of adolescents on ART that have a VL less than 1000 copies/mL at 12 months from study enrolment.
To determine the prevalence of Drug Resistance Mutations(DRMs) among adolescents on ART with a VL≥1000 | 12 months
  Prevalence of DRMs within each drug class will be determined: frequency of single-drug class DRMs vs. dual-class DRMs vs. triple-class DRMs. Frequencies will be assessed for clinically-relevant point mutations to national 1st- and 2nd-line ART regimens

CONTACTS AND LOCATIONS:
Overall Officials: Chiratidzo E NDHLOVU, MD, Principal Investigator — University of Zimbabwe
Locations (1):
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF